CLINICAL TRIAL: NCT02051881
Title: The Identification and Spatial Distribution of Different Nutrient Receptors Along the Gastrointestinal (GI) Tract
Brief Title: Identification of Nutrient Receptors Gastrointestinal Tract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: NL39168.068.12
Record Dates: First submitted 2014-01-30; First posted 2014-01-31 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Distribution of Nutrient Receptors Studied in Intestinal Tissue Obtained Via Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biopsies (Other): Intestinal biopsies were taken in patients who underwent endoscopy.
  Interventions: Other: Taking intestinal biopsies

INTERVENTIONS:
Other: Taking intestinal biopsies

SUMMARY:
Investigating which receptors are involved in nutient sensing of enteroendocrine cells and on nerve endings, gives further knowledge on the kind of nutrients responsible for the secretion of gut hormones involved in satiety signalling. So far only little is know about the distribution of potential nutient sensing receptors along the gastrointestinal tract. The investigators are interested in the intestinal parts which highly secrete CCK and GLP-1. By comparing these tissues, it is expected to further elucidate which receptors are important for satiety signalling in the intestine.

Having this information gives rise to further reseach on how these receptors stimulate the secretion of gut hormones. Moreover, knowing which receptors are involved in satiety signalling, gives oppertunity for targeting these receptors to increase satiety and influencing food intake.

The investigators aim to investigate the distribution of the above mentioned receptors, in the following referred to as 'nutrient sensing receptors', which have been suggested to be involved in satiety signalling, throughout the intestinal tract. For these receptors the gene expression, localisation and protein expression will be determined at different locations. This will be measured in intestinal mucosal biopsies of two locations in the duodenum, in the terminal ileum, the ascending colon, the transverse colon and the descending colon.

ELIGIBILITY:
Inclusion criteria for duodenal biopsies:

* Step 1 (patients asked for participation):

  1. Patients (male and female between 18 and 65 years) referred for upper GI endoscopy (because of functional complaints)
  2. Based on medical history and previous examination, no objection arises for taking extra biopsies during the gastroduodenoscopy.
* Step 2 (patients agreed to participate and in whom biopsies will be taken) 1) Patients with no relevant endoscopic abnormalities (gastroduodenoscopy): patients without gastric or duodenal ulcers/polyps/lesions suspect for malignancy and esophageal lesions or varices.

Inclusion criteria for ileal and colon biopsies:

* Step 1 (patients asked for participation):

Patients (male and female between 18 and 65 years) referred for colonoscopy (because of screening for colorectal cancer or follow up of colonic polyps) Based on medical history and previous examination, no objection arises for taking extra biopsies during the colonoscopy

* Step 2 (patients agreed to participate and in whom biopsies will be taken) Patients with no relevant endoscopic abnormalities (colonoscopy): patients without ileal and/or colonic ulcers/polyps/diverticula and lesions suspect for malignancy Ileum can be reached during colonoscopy

Exclusion criteria for duodenal and ileal colon biopsies:

1. History of severe cardiovascular, gastrointestinal/ hepatic, hematological/immunologic, metabolic/nutritional disease and/or laboratory assessments which might limit participation in the study. The severity of the disease (major interference with the execution of the experiment or potential influence on the study outcomes) will be decided by the principal investigator.
2. Use of medication, which could interfere with normal coagulation (anticoagulants, antiplatelet drugs).
3. Major abdominal surgery interfering with gastrointestinal function (uncomplicated appendectomy, cholecystectomy and hysterectomy allowed, and other surgery upon judgement of the principle investigator)
4. Excessive alcohol consumption (>20 alcoholic consumptions per week)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-05; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Measurements of the expression of receptors with quantitative reverse transcription polymerase chain reaction (q-PCR) in mucosal biopsies of the duodenum, terminal ileum and colon. | 1 day
  Measurements of the expression of receptors with quantitative reverse transcription polymerase chain reaction (q-PCR) in mucosal biopsies of the duodenum, terminal ileum and colon.

SECONDARY OUTCOMES:
Measurements of the location of the receptors with immunohistological techniques in mucosal biopsies of the duodenum, terminal ileum and colon. | 1 day
  Measurements of the location of the receptors with immunohistological techniques in mucosal biopsies of the duodenum, terminal ileum and colon.
Measurements of protein expression in mucosal biopsies of the duodenum, terminal ileum and colon. | 1 day
  Measurements of protein expression in mucosal biopsies of the duodenum, terminal ileum and colon.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Masclee, MD,PhD, Principal Investigator — Maastricht University Medical Center